CLINICAL TRIAL: NCT00119158
Title: An Exploratory Double-blind, Randomized, Vehicle-controlled, Paired Study to Evaluate the Efficacy and Safety of Concomitant Use of Elidel Cream 1% and Cutivate Cream 0.05% in Patients With Severe Lesions of Atopic Dermatitis (AD)
Brief Title: Combination Therapy for Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Jonathan Spergel, The Children's Hospital of Philadelphia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2004-10-3975
Record Dates: First submitted 2005-07-05; First posted 2005-07-13 (Estimated); Results first posted 2010-07-22 (Estimated); Last update posted 2010-07-27 (Estimated); Status verified 2010-07

CONDITIONS: Atopic Dermatitis
Keywords: THerapy for acute moderate to severe flares
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Fluticasone; pimecrolimus

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): Placebo cream
  Interventions: Drug: pimecrolimus
- pimecrolimus cream (Active Comparator)
  Interventions: Drug: Combination of pimecrolimus and fluticasone; Drug: pimecrolimus

INTERVENTIONS:
Drug: Combination of pimecrolimus and fluticasone — Pimecrolimus cream twice a day and fluticasone cream once a day
  Other Names: Pimecrolimus cream; fluticasone
  Arms: pimecrolimus cream
Drug: pimecrolimus — apply daily with fluticasone cream for flares

SUMMARY:
Atopic dermatitis is a chronic relapsing disease with acute flares. The standard therapy is to treat acute flares using topical medications. The two most common classes of topical medications for atopic dermatitis (AD) are topical corticosteroids and topical calcineurin inhibitors.

Pimecrolimus and topical corticosteroids exert their activity by different mechanisms, there may be a synergistic effect of the combination therapy. Therefore, a combination therapy may provide a faster resolution of severe skin lesions and consequently reduce the duration of the topical corticosteroid treatment. Another benefit of the combination therapy maybe the use of a lower potency corticosteroid to achieve the same degree of clearance.

The hypothesis of this trial is that the combination of the two agents will lead to faster clearance than the single agent of topical corticosteroids.

DETAILED DESCRIPTION:
This trial is a double-blind controlled trial of fluticasone cream daily and pimecrolimus cream BID versus fluticasone cream daily and placebo cream BID for the treatment of acute flares of atopic dermatitis.

While pimecrolimus cream 1% has been proven to be effective in mild and moderate Atopic dermatitis (AD), there is a need for a fast control of severe skin lesions. On the other hand, reducing the duration of the topical corticosteroid treatment is a reasonable approach to minimize the occurrence of adverse effects.

Because pimecrolimus and topical corticosteroids exert their activity by different mechanisms, there may be a synergistic effect of the combination therapy. Therefore, a combination therapy may provide a faster resolution of severe skin lesions and consequently reduce the duration of the topical corticosteroid treatment. Another benefit of the combination therapy maybe the use of a lower potency corticosteroid to achieve the same degree of clearance.

In vitro data have demonstrated that a combination of steroids and tacrolimus has synergistic effects on in vitro human lymphocyte proliferation. In addition, it has previously been reported, in a pilot investigation in two subjects, that a combination regimen of pimecrolimus 1% twice a day and fluticasone propionate cream 0.05% once daily was superior to fluticasone propionate cream 0.05% once daily in the acute treatment of atopic dermatitis (AD).

This study is conducted to validate these findings in a larger number of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 2 to 65 years
* Clinical diagnosis of (Atopic Dermatitis) AD according to the American Academy of Dermatology (AAD) Consensus Conference (2001)
* At least two lesions of AD on symmetrical part of the body (same location for each side of the body), of severe intensity (m-EASI is at least 7 on each site, with erythema of at least 3 (severe) and papulation/infiltration of at least 3 (severe)) and similar severity (m-EASI does not differ from more than 2 points on both sides)
* Signed written informed consent
* Willingness and ability to comply with the study requirements
* Female is able to enter and participate in this study if she is of:

  * Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) or
  * Childbearing potential, has a negative pregnancy test (urine) at the screen visit and agrees to an adequate method of birth control throughout the study (which may, at the investigator's discretion, include abstinence)

Exclusion Criteria:

* History of immune deficiencies or history of malignant disease
* Patients with moderate to severe lichenification at the target areas (i.e. score 2 or 3)
* Active cutaneous bacterial, viral or fungal infections in target areas
* History of other skin disorders, including Netherton syndrome, that could interfere with the evaluations
* Use of any topical treatment known or suspected to have an effect on atopic dermatitis within one week prior to the screen visit (except for calcineurin inhibitors, for which the washout is 2 weeks)
* Use of any systemic treatment (including phototherapy) known or suspected to have an effect on AD within four weeks prior to the screen visit [(patients on a stable and low dose of inhaled steroids, on a stable dose of anti histamines, on stable dose of leukotriene antagonists, or receiving occasional short-acting b2-agonists for the treatment of asthma and topical corticosteroids (nasal spray) for the treatment of allergic rhinitis may participate). High-dose inhaled corticosteroids (> 440 mcg of fluticasone a day) and anti-IgE products are not permitted].
* Known sensitivity to pimecrolimus or vehicle (placebo) or fluticasone propionate cream or any of their ingredients
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study
* Use of any other investigational agent in the last 30 days

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2004-10; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan M Spergel, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia
Locations (3):
- United States (3):
  - National Jewish Research Medical Center, Denver, Colorado
  - Northwestern University School of Medicine, Chicago, Illinois
  - University of Texas at Houston Medical School, Houston, Texas

REFERENCES:
- [Background] Spergel J, Hultsch T. Pimecrolimus cream 1% and fluticasone propionate cream 0.05% versus fluticasone propionate cream 0.05% for the treatment of flares of atopic dermatitis. 28th Annual Hawaii Dermatology Seminar, 2004
- [Background] Leung DY, Boguniewicz M, Howell MD, Nomura I, Hamid QA. New insights into atopic dermatitis. J Clin Invest. 2004 Mar;113(5):651-7. doi: 10.1172/JCI21060. PMID 14991059
- [Background] Grassberger M, Baumruker T, Enz A, Hiestand P, Hultsch T, Kalthoff F, Schuler W, Schulz M, Werner FJ, Winiski A, Wolff B, Zenke G. A novel anti-inflammatory drug, SDZ ASM 981, for the treatment of skin diseases: in vitro pharmacology. Br J Dermatol. 1999 Aug;141(2):264-73. doi: 10.1046/j.1365-2133.1999.02974.x. PMID 10468798
- [Background] Eichenfield LF, Lucky AW, Boguniewicz M, Langley RG, Cherill R, Marshall K. 1% pimecrolimus cream for atopic dermatitis. Arch Dermatol. 2003 Oct;139(10):1369-70; author reply 1370-1. doi: 10.1001/archderm.139.10.1369. No abstract available. PMID 14568846
- [Background] Wahn U, Bos JD, Goodfield M, Caputo R, Papp K, Manjra A, Dobozy A, Paul C, Molloy S, Hultsch T, Graeber M, Cherill R, de Prost Y; Flare Reduction in Eczema with Elidel (Children) Multicenter Investigator Study Group. Efficacy and safety of pimecrolimus cream in the long-term management of atopic dermatitis in children. Pediatrics. 2002 Jul;110(1 Pt 1):e2. doi: 10.1542/peds.110.1.e2. PMID 12093983
- [Background] Lee MJ, Pyszczynski N, Jusko WJ. Combined inhibition effects of tacrolimus and methylprednisolone on in vitro human lymphocyte proliferation. Immunopharmacol Immunotoxicol. 1995 May;17(2):335-45. doi: 10.3109/08923979509019755. PMID 7544367
- [Background] Hanifin JM, Thurston M, Omoto M, Cherill R, Tofte SJ, Graeber M. The eczema area and severity index (EASI): assessment of reliability in atopic dermatitis. EASI Evaluator Group. Exp Dermatol. 2001 Feb;10(1):11-8. doi: 10.1034/j.1600-0625.2001.100102.x. PMID 11168575

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical clinics at academic centers
Pre-assignment Details: Patients are self controls. Equivalent areas of eczema were compared
Groups:
- Active Therapy; Placebo Arm: Patients had equivalent eczema on each side of the body. One side of the body was treated with 1% pimecrolimus cream twice a day and fluticasone cream once a day. The opposite side of the body was treated with placebo cream twice a day and fluticasone cream once a day
Period: Active Treatment
Arm/Group | Active Therapy | Placebo Arm
Started | 45 (patients are self controls) | 45
Completed | 45 | 45
Not Completed | 0 | 0
Period: Placebo Treatment
Arm/Group | Active Therapy | Placebo Arm
Started | 45 | 45
Completed | 45 | 45
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Therapy | Placebo Arm | Total
Number analyzed (Participants) | 45 | 45 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 22 | 44
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 16.2 (17.4) | 16.2 (17.4) | 16.2 (17.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 18 | 18 | 36
Region of Enrollment [Number; unit: participants]
  United States | 45 | 45 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the m-EASI (Eczema Area Severity Index) Score.
Description: Eczema Area severity index (EASI) is a composition of scores based on area of eczema involved, (0 = mild to 3 = severe) for four separate Atopic Dermatitis (AD) symptoms: erythema,infiltration ⁄population, excoriation and ichenification.
  Total score 0-12
Time Frame: up to 15 days
Population: Analysis was per protocol, last observation carried forward
Measure: Mean (Standard Deviation); unit: units of a 0-12 scale
Arm/Group | Active Therapy | Placebo Arm
Number analyzed (Participants) | 45 | 45
units of a 0-12 scale | 5.04 (2.7) | 4.77 (2.4)
Statistical Analysis 1: Comparison: Active Therapy; Test type: Non-Inferiority or Equivalence — modified EASI (eczema area severity index) was considered equivalent if p value was greater than >0.05; p < 0.05, t-test, 2 sided

2. Secondary Outcome: The Time to Clearance of the Disease
Description: The time to clearance of eczema measured in days
Time Frame: assessed up to 30 days following drug application
Measure: Mean (Standard Error); unit: days
Arm/Group | Active Therapy | Placebo Arm
Number analyzed (Participants) | 45 | 45
days | 9.22 (4.5) | 7.88 (3.88)

3. Secondary Outcome: The Time to the First Day When m-EASI is Scored by the Investigator as 2 or Less
Description: Time to partial clearance of the localized eczema lesion assessed by the investigator is measured in days
Time Frame: up to one week
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: days

4. Secondary Outcome: The Percentage of Target Areas Reaching a l-IGA (Localized Investigator Global Assessment (l-IGA) or 0 or 1)
Description: The Investigator Global Assessment (IGA) and l-IGA were graded on a scale of 0-4 (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe). The percentage of eczema lesions from the total population that reach almost clear
Time Frame: up to 15 days
Reporting Status: Not Posted
Measure: Mean (Standard Error); unit: percentage of participants

5. Secondary Outcome: The Percentage of Target Areas Improved (i.e., Decrease in Localized Investigator Global Assessmet (l-IGA) Score From Baseline)
Description: The percentage of eczema areas that show improvement in l-IGA score.
  The l-IGA were graded on a scale of 0-4 (0 = clear, 1 = almost clear, 2 = mild disease, 3 = moderate disease, 4 = severe disease).
Time Frame: up to 15 days
Reporting Status: Not Posted
Measure: Mean (Standard Error); unit: percentage of participants

6. Secondary Outcome: The Percentage of Target Areas Reaching a m-EASI (Modifed-Eczema Area Severity Index) Score of 2 or Less
Description: The EASI is a measure of Atopic Dermatitis (AD) severity. A m-EASI score (0-12) was also calculated as the sum of severity (0 = mild to 3 = severe) for four separate AD symptoms: erythema, infiltration ⁄population, excoriation and lichenification.
  The percentage of participants whose eczema reaches almost clear
Time Frame: up to one week
Reporting Status: Not Posted
Measure: Mean (Standard Error); unit: percentage

7. Secondary Outcome: Change From Baseline in Patients' Self Assessment of Disease Severity (PSA) of Target Areas
Description: The patient or caregiver assessment of eczema severity (PSA) was recorded daily in a diary using a 0-4 scale similar to that of the IGA.(0 = clear,
  1 = almost clear, 2 = mild disease, 3 = moderate disease,4 = severe disease).
  Difference in value of PSA from baseline to end of study
Time Frame: 30 days
Reporting Status: Not Posted
Measure: Mean (Standard Error); unit: PSA score of participants

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Active Therapy | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 0/45 | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No